CLINICAL TRIAL: NCT02563405
Title: The Effects of Doxazosin and Nifedipine on Blood Pressure Variability and Uric Acid in Plasma in Hypertensive Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HT-3-UA
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
Keywords: alpha receptor blocker; uric acid; CCB; blood pressure variability
MeSH Terms: conditions — Hypertension | interventions — Doxazosin; Nifedipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxazosin (Active Comparator): To observe the effects of doxazosin (4 mg) on uric acid in plasma and blood pressure variability after 12 weeks of treatment
  Interventions: Drug: Doxazosin; Drug: Nifedipine
- nifedipine (Active Comparator): To observe the effects of nifedipine (30 mg) on uric acid in plasma and blood pressure variability after 12 weeks of treatment
  Interventions: Drug: Doxazosin; Drug: Nifedipine

INTERVENTIONS:
Drug: Doxazosin — Doxazosin was given orally in a dose of 4 mg/day to treat patients in the doxazosin group for 12 weeks.
Drug: Nifedipine — Nifedipine was given orally in a dose of 30 mg/day to treat patients in the amlodipine group for 12 weeks.

SUMMARY:
Hypertension is one of the most common cardiovascular diseases, which is a major risk factor for stroke and cardiovascular events. Accumulated data has shown that target-organ damage is related not only to 24-h mean intra-arterial BP, but also to BP variability (BPV) in subjects with essential hypertension. There are many studies about the effects of different kinds of drugs on blood pressure, but the clinical researches about the impacts of antihypertensive drugs on BPV are limited, and the conclusion is still controversial.

In addition, recent studies found that the occurrence and development of hypertension, especially essential hypertension, are closely related with hyperuricemia. Serum UA is an independently prognostic indicator for the development of hypertension. Some studies have observed the effects of different kinds of antihypertensive drugs on uric acid level in hypertensive patients. After adjustment, calcium channel blockers are associated with a lower risk of incident gout among people with hypertension. However, the effects of alpha blockers on uric acid in plasma are still not very clear.

Therefore, we performed this study to observe the different effects of alpha blocker and calcium channel blocker on blood pressure variability and uric acid level in hypertensive patients.

DETAILED DESCRIPTION:
Hypertension is one of the most common cardiovascular diseases, which is a major risk factor for stroke and cardiovascular events. Traditionally, cardiovascular risk stratification in hypertensive patients was based on the average blood pressure (BP) measured in the clinic. Accumulated data has shown that target-organ damage is related not only to 24-h mean intra-arterial BP, but also to BP variability (BPV) in subjects with essential hypertension. Growing evidence demonstrated that BPV has considerable prognostic value for all-cause mortality and cardiovascular outcomes, independent of average BP. At present, the normal range of BPV is not very clear. There are many studies about the effects of different kinds of drugs on blood pressure, but the clinical researches about the impacts of antihypertensive drugs on BPV are limited, and the conclusion is still controversial.

In addition, recent studies found that the occurrence and development of hypertension, especially essential hypertension, are closely related with hyperuricemia. Accumulated data has shown that a significant and independent association between the uric acid level and the onset of hypertension in both men and women participants. Serum UA is an independently prognostic indicator for the development of hypertension. Some studies have observed the effects of different kinds of antihypertensive drugs on uric acid level in hypertensive patients. After adjustment, diuretics, β blockers, angiotensin converting enzyme inhibitors and non-losartan angiotensin Ⅱ receptor antagonists are associated with an increased risk of gout. In contrast, calcium channel blockers and losartan are associated with a lower risk of incident gout among people with hypertension. However, the effects of alpha blockers on uric acid in plasma are still not very clear.

Therefore, we performed this study to observe the different effects of alpha blocker and calcium channel blocker on blood pressure variability and uric acid level in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

Men aged between 18 and 75 included years old Postmenopausal women who are no more than 75 years older. Patients with essential mild to moderate uncomplicated hypertension (DBP<110mmHg and SBP<180mmHg measured with a validated automatic device in sitting position) after initiation or intensification of appropriate healthy lifestyle modification, Without antihypertensive treatment in 2 weeks.

Exclusion Criteria:

History of cerebrovascular disease: ischemic stroke, cerebral haemorrhage and TIA.

History of cardiovascular disease:unstable angina, myocardial infarction, coronary revascularization and congestive heart failure.

History of renal impairment. History of Type I diabetes mellitus or Type II diabetes uncontrolled. History of liver impairment. History of alcoholism or drug abuse. Known symptomatic orthostatic hypotension. Contra-indications to treatment with investigate products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
24-hour Ambulatory Blood Pressure Monitoring | 3 years

SECONDARY OUTCOMES:
plasma uric acid level | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- uric acid test and 24-hour ambulatory BP monitoring, Harbin, Heilongjiang, China